CLINICAL TRIAL: NCT00323804
Title: Randomized, Double-blind, Placebo-controlled Multicenter Study Evaluating the Interest of a Long-term (3 Years) Treatment With Peginterferon Alfa-2b and Ribavirin on Liver Fibrosis in Non-responder Chronic Hepatitis C Patients.
Brief Title: Interest of Ribavirin in the Maintenance Treatment of Liver Fibrosis Using Low Dose Pegylated Interferon alpha2b in Patients With Chronic Hepatitis C Non Responders to Previous Antiviral Therapy.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANRS HC15 NRfi; 2005-002937-11 (EudraCT Number)
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-08

CONDITIONS: Hepatitis C, Chronic; Liver Fibrosis
Keywords: Maintenance therapy; Non-responder patients; Ribavirin/peginterferon combination therapy; Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Randomised PegIFN alfa 2b + ribavirin (RBV) arm (Experimental): Combination of ribavirin capsules 200 mg, weight-based daily dose ( <75 kg : 1000 mg ; ≥ 75 kg : 1200 mg), and low-dose PegIFN alfa 2b by subcutaneous injection 0.5 μg / kg / week, from day 0 to M36
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin
- Randomised PegIFN alfa 2b + ribavirin-placebo arm (Placebo Comparator): Combination of ribavirin-placebo capsules 200 mg, weight-based daily dose ( <75 kg : 1000 mg ; ≥ 75 kg : 1200 mg), and low-dose PegIFN alfa 2b by subcutaneous injection 0.5 μg / kg / week, from day 0 to M36
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin-Placebo

INTERVENTIONS:
Biological: Peginterferon alfa-2b — PegIFN alfa 2b in addition to ribavirin or ribavirin-placebo, from day 0 to M36
Drug: Ribavirin — Ribavirin in addition to PegIFN alfa 2b, from day 0 to M36
  Arms: Randomised PegIFN alfa 2b + ribavirin (RBV) arm
Drug: Ribavirin-Placebo — Ribavirin-placebo in addition to PegIFN alfa 2b, from day 0 to M36
  Arms: Randomised PegIFN alfa 2b + ribavirin-placebo arm

SUMMARY:
Patients with chronic hepatitis C who did not respond to previous antiviral treatment develop liver fibrosis leading to cirrhosis. Maintenance low dose pegylated interferon therapy of fibrosis is currently under investigation in large multicenter trials. The aim of our study is to assess if peginterferon alpha2b plus ribavirin is more efficient than peginterferon alpha2b alone. 454 patients will be randomized between the 2 arms and the efficacy will be assessed, after 3 years of treatment, on Metavir liver fibrosis score improvement.

DETAILED DESCRIPTION:
Up to 45% of patients with chronic hepatitis C do not respond to pegylated interferon/ribavirin combination therapy. These patients are prone to develop liver fibrosis leading to cirrhosis and its complications. Interferon has proven to be efficient in liver fibrosis treatment even in case of virological non response. Maintenance low dose pegylated interferon therapy is currently under investigation in large multicenter trials. The aim of our study is to assess wether peginterferon alpha 2 b (0.5 µg/kg/week) plus ribavirin (800-1200 mg according to body weight) is more efficient than peginterferon alpha 2 b alone in a long term 3 years treatment of liver fibrosis. 454 patients, non responders (VHC RNA positive after 24 weeks of treatment or absence of ≥ 2 log HCV RNA drop after 12 weeks of treatment) to a previous peginterferon/ribavirin antiviral treatment will be randomized between the 2 arms, with a double-blind masking of ribavirin. The efficacy will be assessed on Metavir liver fibrosis score improvement between pre and post therapeutic liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18
* With a hepatitis C virus infection (HCV RNA and anti-HCV antibodies in serum)
* Not responders to a previous antiviral treatment using the interferon plus ribavirin combination
* With a wash-out of treatment for at least 6 months
* With an active chronic hepatitis C and a Metavir fibrosis score ≥ 2
* Serum ALT levels > upper limit of the laboratory on two occasions within 6 months before inclusion
* Accepting to undergo a liver biopsy at the end of the study
* Negative pregnancy test for women
* With a social security cover
* Written informed consent

Exclusion Criteria:

* History of hepatic complications
* History of transplantation
* History of severe seizures
* History of severe psychiatric disorders
* Drug addiction within the last 12 months
* Associated condition susceptible to be responsible for liver fibrosis
* Hepatocellular carcinoma
* Cardiovascular disease unstable under treatment
* Uncontrolled diabetes
* Retinopathy
* Thyroid disease unstable under treatment
* Epilepsy and/or central nervous system functional disorders
* Autoimmune disease
* Regular alcohol consumption
* Pregnancy, breast-feeding or absence of contraception
* Haemoglobin <12 g/dl
* platelets <50000/mm3
* Neutrophils < 1200/ mm3
* Severe hepatocellular failure (prothrombin index lower than 60%)
* Renal failure (creatinine clearance lower than 50 mL/Mn)
* Associated immunosuppressive drugs, corticosteroids, antiviral drugs (other than study ones)
* Treatment with drugs likely to have an effect on fibrosis
* Anticonvulsants
* Inability to tolerate interferon

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2006-05; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Rate of patients with at least a one point improvement in Metavir fibrosis score between the inclusion and the end-of-study liver biopsies. | Screen visit and M36

SECONDARY OUTCOMES:
Distribution of the Metavir scoring on the end-of-study biopsy | M36
Distribution of the Chevallier fibrosis score | Screen visit and M36
Evolution of the area of fibrosis between the inclusion and the end-of -study biopsies | Screen visit and M36
Fibrosis serum markers | Screen, day0, M6, M12, M24, M36
Liver elasticity before and after treatment | Screen,M12, M24, M36
Safety of treatment and quality of life | day0, M6, M12, M24, M36
Frequency of occurrence of hepatic complications and/or liver transplantations | Day 0 to M36
Evolution of the hepatitis C viral load | Screen to M36
Rate of patients with loss of detectable hepatitis C virus RNA | Day 0 to M36

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Guyader, MD, PhD, Principal Investigator — CHU Rennes; Eric Bellissant, MD, PhD, Study Chair — CHU Rennes
Locations (45):
- Belgium (5):
  - CHU Brugmann, Brussels
  - Hôpital Bracops, Brussels
  - Hôpital Erasme, Brussels
  - Hôpital de Jolimont, La Louvière
  - CHU Sart Tilman, Liège
- France (40):
  - Service d'Hépatogastroentérologie et d'endoscopie digestive - CH du Pays d'Aix, Aix-en-Provence
  - Hôpital Nord, Amiens
  - Service d'Hépatogastroentérologie - Hôpital Nord, Amiens
  - Service d'Hépatologie - Gastroentérologie - Cancérologie digestive - CHU Angers, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Service d'Hépatogastroentérologie - Hôpital Avicenne, Bobigny
  - Service d' Hépatogastroentérologie - Hôpital Jean Verdier, Bondy
  - Service d'Hépatogastroentérologie et d'Assistance nutritive - Hôpital Haut-Lévêque, Bordeaux Pessac
  - CH Pierre OUDOT, Bourgoin
  - Service d'Hépatogastroentérologie - Hôpital de la Cavale Blanche, Brest
  - Service d'Hépatologie - Gastroentérologie - Nutrition -Hôpital de la Côte de Nacre, Caen
  - Centre Hospitalier, Châteauroux
  - Service d'Hépatogastroentérologie - CHU d'ESTAING, Clermont-Ferrand
  - Service d'Hépatogastroentérologie - Hôpital Beaujon, Clichy
  - Service d'Hépatogastroentérologie - CH Sud Francilien, Corbeil-Essonnes
  - Service d'Hépatogastroentérologie - Hôpital du Bocage, Dijon
  - Hôpital Nord, Grenoble
  - Service d'Hépatogastroentérologie - CH La Roche sur Yon, La Roche-sur-Yon
  - Service des Maladies du Foie et de l'appareil Digestif - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Département d'Hépatogastroentérologie - CH Le Mans, Le Mans
  - Service d'Hépatogastroentérologie - CHRU - Hôpital Claude Huriez, Lille
  - Service d'Hépatogastroentérologie - Hotel de la Croix Rousse, Lyon
  - Service d'Hépatogastroentérologie - Hôpital Saint Joseph, Marseille
  - Service d'Hépatogastroentérologie - CH Montauban, Montauban
  - Service d'Hépatogastroentérologie - CH Montélimar, Montélimar
  - Service d'Hépatogastroentérologie - Hôpital Saint Eloi, Montpellier
  - Service d'Hépatogastroentérologie - Hôtel Dieu, Nantes
  - Hôpital de l'Archet, Nice
  - Service d'Hépatogastroentérologie - Hôpital de la Source, Orléans
  - Service d'Hépatogastroentérologie - Hôpital La Pitié Salpétrière, Paris
  - Service d'Hépatogastroentérologie - Hôpital Tenon, Paris
  - Service d'Hépatogastroentérologie - Hôpital Pontchaillou, Rennes
  - Service d'Hépatogastroentérologie - CHU Rouen, Rouen
  - Centre Hospitalier, Saint-Quentin
  - Service d'Hépatogastroentérologie, Clinique médicale B - Hôpital Civil, Strasbourg
  - Hôpital Purpan, Toulouse
  - Service d'Hépatogastroentérologie - Hôpital Purpan, Toulouse
  - Service d'Hépatogastroentérologie - Hôpital Trousseau, Tours
  - Service d'Hépatogastroentérologie - Hôpital Brabois, Vandœuvre-lès-Nancy
  - Hôpita Paul Brousse, Villejuif